CLINICAL TRIAL: NCT05215769
Title: Video Intervention to Address Pre-Test Patient Education for Tumor Genomic Testing
Brief Title: A Video Intervention to Improve Patient Understanding of Tumor Genomic Testing in Patients With Metastatic Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Daniel Stover, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: OSU-21313; NCI-2021-13900 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); R21CA259985 (NIH)
Record Dates: First submitted 2022-01-18; First posted 2022-01-31 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Anatomic Stage IV Breast Cancer AJCC v8; Metastatic Breast Carcinoma; Metastatic Lung Carcinoma; Metastatic Malignant Solid Neoplasm; Prognostic Stage IV Breast Cancer AJCC v8; Stage IV Lung Cancer AJCC v8; Stage IVA Lung Cancer AJCC v8; Stage IVB Lung Cancer AJCC v8
MeSH Terms: conditions — Breast Neoplasms; Lung Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Health services research (video) (Experimental): Patients participate in a video intervention session and complete questionnaires at baseline, after participating in the video intervention, and after receiving NGS results.
  Interventions: Behavioral: Health Education; Other: Questionnaire Administration

INTERVENTIONS:
Behavioral: Health Education — Participate in a video intervention
Other: Questionnaire Administration — Complete questionnaires

SUMMARY:
This clinical trial tests whether a video intervention improves patient understanding of tumor genomic testing in patients with cancer that has spread to other parts of the body (metastatic). Measuring how the video intervention affects patient understanding of tumor genomic testing in patients with metastatic cancer may help doctors provide patient-centered care by effectively communicating the importance of tumor genomic testing.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess change in patient knowledge about tumor next generation sequencing (NGS) following exposure to the video.

SECONDARY OBJECTIVES:

I.To assess changes following exposure to the video, including; Ia. Genomic knowledge via the validated 10 true/false question survey (% correct out of 10).

Ib. 11-item Trust in Physician Survey (TPS) as a single TPS score. Ic. Comparison of results in three patient cohorts: 1) Metastatic breast cancer; 2) lung cancer; 3) metastatic cancer of unspecified type.

EXPLORATORY OBJECTIVE:

I. Assess whether therapies prescribed as a result of tumor NGS achieved clinically favorable result through chart review.

OUTLINE:

Patients participate in a video intervention session and complete questionnaires at baseline, after participating in the video intervention, and after receiving NGS results.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have biopsy-confirmed metastatic cancer
* Be >= 18 years of age
* Be undergoing clinical tumor or circulating tumor deoxyribonucleic acid (DNA) NGS

Exclusion Criteria:

* Exclude patients who are not English- or Spanish-speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 243 (Actual)
Dates: Start 2022-03-30 (Actual); Primary Completion 2025-01-27 (Actual); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Message-specific knowledge/recall accuracy | Immediately before and immediately after video intervention
  Measured as number correct out of 10 questions. Will have 90% power to detect an effect size of 0.47 in change of recall accuracy from pre- to post- video intervention, using a two-sided Wilcoxon signed-rank test with alpha of 0.05.

SECONDARY OUTCOMES:
Change in patient genomic knowledge | Immediately before and immediately after video intervention
  Measured with the validated 10 true/false question survey (% correct out of 10). Will be summarized using descriptive statistics and compared pre-/post-video using Wilcoxon signed rank test.
Change in patient trust of physician/provider | Immediately before and immediately after video intervention
  Measured with the 11-item trust in physician survey (TPS) as a single TPS score. Will be summarized using descriptive statistics and compared pre-/post-video using Wilcoxon signed rank test.
Change in patient genomic knowledge in metastatic breast cancer (MBC) versus metastatic lung cancer (MLC) patients | Immediately before and immediately after video intervention
  Measured with the validated 10 true/false question survey (% correct out of 10). Will be summarized using descriptive statistics and compared pre-/post-video using Wilcoxon signed rank test. Will be compared between MBC and MLC patients using Wilcoxon rank sum test.
Change in patient trust of physician/provider in MBC versus MLC patients | Immediately before and immediately after video intervention
  Measured with the 11-item TPS as a single TPS score. Will be summarized using descriptive statistics and compared pre-/post-video using Wilcoxon signed rank test. Will be compared between MBC and MLC patients using Wilcoxon rank sum test.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel G Stover, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (4):
- United States (4):
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - St. Rita's, Lima, Ohio
  - Saint Francis Medical Center, Richmond, Ohio
  - Saint Elizabeth Youngstown Hospital, Youngstown, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Veney D, Wei L, Toland AE, Presley CJ, Hampel H, Padamsee TJ, Lee CN, Irvin WJ Jr, Bishop M, Kim J, Hovick SR, Senter L, Stover DG. A Video Intervention to Improve Patient Understanding of Tumor Genomic Testing in Patients with Cancer. medRxiv [Preprint]. 2023 Dec 5:2023.12.05.23299443. doi: 10.1101/2023.12.05.23299443. PMID 38106014
- See also: The Jamesline — http://cancer.osu.edu